CLINICAL TRIAL: NCT03180138
Title: Enhancing Health Care Access With Cellular Technology: Networked and Mobile Technologies to Improve Uptake and Coverage of Vaccinations
Brief Title: Enhancing Health Care Access With Cellular Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Ministry of Science and Technology, India (Other Government); Bal Umang Drishya Sanstha (BUDS), India (Other); Royal Datamatics Pvt. Ltd. (RDPL), India (Unknown); St. Louis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00086292; R03EB015955 (NIH)
Record Dates: First submitted 2017-06-05; First posted 2017-06-08 (Actual); Results first posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Vaccination
Keywords: mobile phone; Children's Health

STUDY DESIGN:
Intervention Model Description: Single blinded prospective study
Who Masked: Investigator
Masking Description: Study team members are blinded to group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Controls (No Intervention)
- Reminders alone (Active Comparator)
  Interventions: Behavioral: Reminders alone
- Reminders + compliance-linked incentives (Active Comparator)
  Interventions: Behavioral: Reminders alone; Behavioral: Compliance-linked incentives

INTERVENTIONS:
Behavioral: Reminders alone — Automated reminders (text and /or voice in local language) for upcoming vaccination visit(s) will be provided via cell-phone to the subject (mother / caregiver) or pregnant woman.
  Arms: Reminders + compliance-linked incentives; Reminders alone
Behavioral: Compliance-linked incentives — Automated compliance-linked incentives (as cell-phone minutes) will be provided via cell-phone to the subject (mother / caregiver) or pregnant woman.
  Arms: Reminders + compliance-linked incentives

SUMMARY:
Despite the impressive economic progress in developing countries, significant proportion of young children and pregnant women living in low-resource settings remain inadequately immunized. Progressive decline in immunizations are in large part attributable to poor follow-up and compliance. National and international pediatric bodies, recommend a time sensitive schedule for childhood immunizations, boosting immunity with each subsequent cycle, leading to adequate levels of immune protection. Due to inadequate protective immunity, resulting from poor vaccination compliance, outbreaks of vaccine-preventable diseases are rampant, making childhood mortality in this group among the highest in the world. Major challenges of vaccination programs include maintaining / tracking records, linked to positive identification of individual children, and strategies to improve follow-up and compliance. Novel cellular technology based approaches targeting behavior modifications can therefore significantly impact health outcomes in these communities. In this proposal, the investigators will evaluate a novel software platform, utilizing biometric identification of subjects, paired with cell-phone reminders and compliance-linked incentives to improve uptake and coverage of primary vaccinations in young children and pregnant women.

DETAILED DESCRIPTION:
A web-based, biometric-linked vaccination record, cell-phone reminder and compliance-linked incentive software platform to provide robust and universal access of vaccinations. The investigators will implement this platform in a low-resource settings with the following features: a) Web-based for robust and universal access. b) Biometric-linked for positive identification. c) Digital storage and reporting for transparent view of program operations. d) Global Positioning System (GPS)-linked, allowing rapid assessment of vaccination status of communities. e) Increasing vaccination uptake and coverage by automated text message reminders and compliance-linked incentives.

ELIGIBILITY:
Inclusion Criteria:

Mother-child (or caregiver-child) units with child <2 years of age OR Pregnant women

Exclusion Criteria:

Family does not have cell-phone OR cannot provide informed consent

Max Age: 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 608 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay K Jain, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276
- [Derived] Seth R, Akinboyo I, Chhabra A, Qaiyum Y, Shet A, Gupte N, Jain AK, Jain SK. Mobile Phone Incentives for Childhood Immunizations in Rural India. Pediatrics. 2018 Apr;141(4):e20173455. doi: 10.1542/peds.2017-3455. Epub 2018 Mar 14. PMID 29540571

RESULTS

PARTICIPANT FLOW:
Groups:
- Controls: A cloud-based, biometric-linked software platform was used for positive identification, and record keeping.
- Reminders Alone: Reminders alone: Automated reminders (text and /or voice in local language) for upcoming vaccination visit(s) will be provided via cell-phone to the subject (mother / caregiver).
  A cloud-based, biometric-linked software platform was used for positive identification, and record keeping.
- Reminders + Compliance-linked Incentives: Reminders alone: Automated reminders (text and /or voice in local language) for upcoming vaccination visit(s) will be provided via cell-phone to the subject (mother / caregiver).
  Compliance-linked incentives: Automated compliance-linked incentives (as cell-phone minutes) will be provided via cell-phone to the subject (mother / caregiver).
  A cloud-based, biometric-linked software platform was used for positive identification, and record keeping.
Period: Overall Study
Arm/Group | Controls | Reminders Alone | Reminders + Compliance-linked Incentives
Started | 204 | 201 | 203
Completed | 182 | 188 | 179
Not Completed | 22 | 13 | 24
Not completed — Mobile-phone could not be verified | 2 | 13 | 15
Not completed — No prior immunization records | 17 | 0 | 6
Not completed — Found to be >24 mon after randomization | 3 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Controls | Reminders Alone | Reminders + Compliance-linked Incentives | Total
Number analyzed (Participants) | 182 | 188 | 179 | 549
Age, Continuous [Median (Inter-Quartile Range); unit: Months] | 5 [1 to 11] | 5 [1 to 11] | 4 [1 to 11] | 5 [1 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 97 | 90 | 282
  Male | 87 | 91 | 89 | 267
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 182 | 188 | 179 | 549
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Immunization Rate
Description: Percent of the total number of immunizations received divided by the total number of immunizations required at the time of measurement for each child. Calculated for each child and in each cohort.
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: Percentage of immunizations
Arm/Group | Controls | Reminders Alone | Reminders + Compliance-linked Incentives
Number analyzed (Participants) | 182 | 188 | 179
Percentage of immunizations | 41.7 [23.1 to 69.2] | 40.1 [30.8 to 69.2] | 50.0 [30.8 to 76.9]

2. Secondary Outcome: Timeliness of Vaccinations
Description: The percent of immunizations administered before or within 14 days after the scheduled date for the immunization. Calculated for each cohort.
Time Frame: 12 months
Population: The events analyzed here are the total number of vaccines rather than subjects in each cohort. The outcome measure is the percent of the number of vaccines that were administrated in a timely manner divided by the total number of scheduled vaccines.
Measure: Number; unit: Percentage of vaccines
Units Other Than Participants: Vaccines
Arm/Group | Controls | Reminders Alone | Reminders + Compliance-linked Incentives
Number analyzed (Participants) | 182 | 188 | 179
Number analyzed (Vaccines) | 243 | 243 | 287
Percentage of vaccines | 31.6 | 24.7 | 40.8

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Controls | Reminders Alone | Reminders + Compliance-linked Incentives
All-Cause Mortality (participants affected / at risk) | 0/182 | 0/188 | 0/179
Serious Adverse Events (participants affected / at risk) | 0/182 | 0/188 | 0/179
Other Adverse Events (participants affected / at risk) | 0/182 | 0/188 | 0/179

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT03180138/Prot_SAP_000.pdf